CLINICAL TRIAL: NCT07187414
Title: Microbiological Description of Sperm and Follicular Fluid Samples. Impact on IVF/ICSI Success Rates (SPERMIBIOTE)
Brief Title: Microbiological Description of Sperm and Follicular Fluid Samples. Impact on IVF/ICSI Success Rates
Acronym: SPERMIBIOTE
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-06-044-ERAMO0574
Record Dates: First submitted 2025-09-18; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: In Vitro Fertilization (IVF); Medically Assisted Procreation (MAP)
Keywords: In Vitro Fertilization (IVF); Medically Assisted Procreation (MAP); intracytoplasmic sperm injection (ICSI); microbiota

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The samples analyzed come from the bacteria contained in the culture medium
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to quantify and identify bacteria that may be present in semen and follicular fluid samples on the day of the IVF-ICSI attempt.

The secondary objective is to :

* Quantify and identify bacteria that may be present in embryo culture media on day 6.
* Correlate microbiological analyses of sperm and follicular fluids with those of embryo culture media on day 6.
* Evaluate their impact on fertilization and blastulation rates

DETAILED DESCRIPTION:
This is a single-center observational study based on data contained in the medical records of couples treated and evaluated as part of Medically Assisted Procreation (IVF-ICSI).

This study was conducted at the Parly 2 private hospital for data and sample collection, at the Parly 2 hospital microbiology laboratory, and at Life & Soft Fontenay-aux-Roses for sample analysis.

Collected samples will not be stored after analysis. The objective of this study does not impose any particular constraints. The study consists of a single assessment, the data from which will be recorded on an electronic case report form (CRF).

ELIGIBILITY:
Inclusion Criteria:

* Man aged 18 to 59 who have provided a sperm sample after an abstinence period of between 2 and 7 days. Sperm prepared by density gradient on day 0. Negative sperm culture (<6 months). No specific urogenital history (varicocele, cryptorchidism, testicular ectopia, etc.).
* Women aged 18 to 43 undergoing oocyte puncture with collection of follicular fluid on day 0. No endometriosis or hydrosalpinx. Negative vaginal sample (< 6 months).
* Negative HIV, HBV, and HCV serology tests within the last year.
* Absence of urinary tract infections in men and sexually transmitted infections (HPV, HSV, HIV-1/2, C. trachomatis, Gonorrhea, Syphilis, etc.) (<6 months).
* Absence of recent antibiotic or antifungal treatment (end of treatment < 3 months) Absence of probiotic intake (< 3 months).
* No history of chemotherapy or radiation therapy.
* Embryonic culture performed up to day 6 for all zygotes.

Exclusion Criteria:

* Homosexual patient couples or transsexual couples
* Patients treated for medically assisted procreation with a third-party donor
* Frozen sperm pellets (ejaculate or surgical)
* Donor sperm
* Sperm prepared by washing
* Abstinence period <2 or >7 days
* Fever <3 months
* History of chemotherapy or radiotherapy.
* History of urinary tract infections in man (< 6 months)
* History of sexually transmitted infections (HPV, HSV, HIV-1/2, C. trachomatis, gonorrhea, syphilis, etc.) (<6 months)
* Specific urogenital history (varicocele, cryptorchidism, testicular ectopia, etc.)
* Recent antibiotic therapy or antifungal treatment (end of treatment < 3 months)
* Taking probiotics (end of treatment < 3 months)
* Positive sperm culture < 6 months.
* Positive vaginal sample < 6 months. White puncture.
* Collection failure.
* Fertilization failure

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Collection of data from medical records and analysis of biological samples taken from couples as part of medically assisted procreation care.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-03-29 (Actual); Study Completion 2025-03-29 (Actual)

PRIMARY OUTCOMES:
Quantification and identification of bacteria present in semen and follicular fluid samples on the day of the IVF-ICSI attempt. | Day 0
  Analysis of sequences of bacteria identified by amplification and sequencing of the gene encoding 16S rRNA in aliquots taken on day 0.

SECONDARY OUTCOMES:
Quantification and identification of bacteria present in semen and follicular fluid samples on the day 6 after of the IVF-ICSI attempt. | Day 6
  Description: Analysis of sequences of bacteria identified by amplification and sequencing of the gene encoding 16S rRNA in aliquots taken on day 6.
IVF/ICSI success rate | Day 6
  presence of a morula on day 6

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé de Parly II, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No